CLINICAL TRIAL: NCT03333005
Title: An Open Label, Multi-Center Study to Determine the Safety and Pharmacokinetics of Intravenous and Oral APX001 in Patients Undergoing Chemotherapy for Acute Myeloid Leukemia With Neutropenia
Brief Title: Safety and Pharmacokinetics of Intravenous and Oral APX001 in Patients With Acute Myeloid Leukemia (AML) and Neutropenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: The Clinical Trials Centre Cologne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: APX001-103
Record Dates: First submitted 2017-10-23; First posted 2017-11-06 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: The first 10 patients enrolled will be administered IV APX001. The second 10 patients enrolled will be administered oral APX001
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APX001 with Standard of Care Anti-fungal agent (Experimental)
  Interventions: Drug: APX001 with Standard of Care anti-fungal agent

INTERVENTIONS:
Drug: APX001 with Standard of Care anti-fungal agent — safety assessment

SUMMARY:
An open-label, multi-center, Phase Ib study to determine the safety and pharmacokinetics of intravenous and oral APX001 in patients undergoing chemotherapy for Acute Myeloid Leukemia with neutropenia.

A total of 20 patients will be enrolled in this study. 10 patients in Cohort I, intravenous drug dosing and 10 patients will be enrolled in Cohort II, oral drug dosing.

All patients will receive chemotherapy for their AML according to local clinical standard of care as well as antifungal prophylaxis.

APX001 will be administered for 14 consecutive days, beginning on Study Day 3 after onset of chemotherapy

ELIGIBILITY:
Key Inclusion Criteria:

* Provision of written consent
* Ages 18-75 inclusive, male or female
* Diagnosis of Acute Myeloid Leukemia
* Patients entering first induction treatment chemotherapy
* Expected to be neutropenic (<500 ANC/ul) for >/= 10 days

Key Exclusion Criteria:

* Patients who received systemic antifungal therapy for proven or probable fungal infections within the last 12 months
* Current fever (> 38 degrees Celsius)
* Concomitant use of rifampin, rifabutin, ergot alkaloids, terfenadine, astemizole, cisapride, pimozide, quinidine, long acting barbiturates, neostigmine and carbamazepine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse events as assessed and reported by CTCAE v4.0 | One to forty-four days

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | One to forty-four days
Peak Plasma Concentration (Cmax) | One to forty-four days

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (3):
- Germany (3):
  - University of Cologne, Center for Integrated Oncology (CIO), Cologne
  - Johannes Gutenberg, University of Mainz, Mainz
  - University of Munich, Grosshadern Campus, Munich